CLINICAL TRIAL: NCT05667831
Title: Comparison of the Effects of Two Different Wound Dressing on the Pressure Injury Patients in Long-term Care Institutions
Brief Title: The Effects of Alginate Ag Dressing in the Pressure Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Shu-Fen Lo, Associate Professor, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC110-27
Record Dates: First submitted 2022-06-03; First posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Pressure Injury; Long-Term Care
Keywords: pressure injury; patient; wound infection; nurses
MeSH Terms: conditions — Pressure Ulcer; Wound Infection

STUDY DESIGN:
Intervention Model Description: Subjects who meet the inclusion criteria of this study will be randomly assigned by the research assistant to the experimental group or the control group by generating random numbers on the computer.
Who Masked: Participant, Care Provider
Masking Description: Before the subjects were assigned, neither the participants, nurses nor the researchers knew whether the subjects were in the experimental group or the control group. When the patients met the inclusion criteria, the research assistant informed the clinical nurses of the results of the case assignment(experimental group or control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alginate silver dressing (Experimental): The experimental group received alginate calcium and silver ion dressing
  Interventions: Other: Alginate silver silver ion dressing
- traditional dressing (No Intervention): Study subjects received traditional dressing changes such as wet dressing or SSD

INTERVENTIONS:
Other: Alginate silver silver ion dressing — Alginate silver silver ion dressing is a soft, comfortable wound dressing with a high mannuronic acid content. Gels on contact with wound exudate or blood, creating a moist wound environment for optimal wound healing. Silver ions protect the dressing from a range of microorganisms.
  Arms: Alginate silver dressing

SUMMARY:
Wound infection and bleeding is a risk factor for pressure injury. Calcium alginate silver dressing (CASD) has been shown to be beneficial in a variety of wounds. However, evidence of its benefit in pressure injury(PI) patients in long-term care institutions, especially with respect to Taiwan population, is sparse. This study was to evaluate the effect of CASD and conventional wound dressings on the PI patients in long-term care institutions.

DETAILED DESCRIPTION:
Background: Wound infection and bleeding is a risk factor for pressure injury. Calcium alginate silver dressing (CASD) has been shown to be beneficial in a variety of wounds. However, evidence of its benefit in PI patients in long-term care institutions, especially with respect to Taiwan population, is sparse.

Objective: To evaluate the effect of CASD and conventional wound dressings on the PI patients in long-term care institutions. The study hypothesis that when using the CASD will improving wound bed status more than conventional dressing change.

Design: Prospective, randomized trial Setting: Multiple center long-term care institutions in Taiwan. Methods: In this clinical trial, 200 PI patients will randomly assigned to treatment with either calcium alginate silver dressing or conventional wound dressings for up to 14 days or to the point of full reepithelialization of the wound. The length and depth of the studied wounds were recorded once a week. The instruments will using the PI measurement tool measured on day0, day7 and day14.The collected data were analyzed by descriptive and inferential statistical methods . The Mann-Whitney test was applied to compare primary endpoint between groups. Differences in secondary endpoint were also compared.

Expected results: PI is an indicator of care quality in long-term care institutions. However, as the population ages, PI are prone to infection and bleeding problems, causing patients to have potential health problems such as sepsis and hemoglobin reduction. The results of this study will provide evidence-based care for wound dressing in long-term care institutions, thereby improving patient care.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20-90 years old
2. Stage II or stage III pressure injury
3. Pressure injury wound size: length, width and depth are less than 10*10*2 cm
4. The patient or family agree to be willing to participate in and cooperate with the interventional treatment of this study

Exclusion Criteria:

1. The wound has a underming wound or a tunnel wound
2. Black crust on the wound bed
3. Participant's with unstable vital signs
4. Those who have used silver dressings or silver hydrofiber dressings in the past 30 days
5. The patient has any other related disease symptoms that may interfere with the safety and efficacy of the study results
6. Long-term care institutions are protected resettlement or homeless people without legal representatives

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change bacterial colony count in wound bed Bacterial colony count in wound bed Bacterial colony count in wound bed | Change from baseline bacterial colony count in wound bed at 14 days
  Take bacteria from the wound bed for wound culture
Change white blood cell count | Change from white blood cell count at 14 day
  Draw 2cc of blood for analysis of white blood cell count
Change high sensitivity C- reactive protein(hsCRP) | Change from hsCRP at 14 day
  Draw 2cc of blood for analysis of white blood cell count

SECONDARY OUTCOMES:
Change Wound Bed Condition Assessment Scale | Change from wound bed condition assessment at 14 day
  The Wound Bed Condition Assessment(WBCA) scale comprised of 8 items rated on a five-point Likert-type scale. The WBCA had a range of possible scores from 8 to 40. A higher score indicated more worse wound bed condition.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen LO, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
According the guidelines of the Declaration of Helsinki.The data presented in this study are available on request from the corresponding author

REFERENCES:
- [Background] Anthony D, Alosoumi D, Safari R. Prevalence of pressure ulcers in long-term care: a global review. J Wound Care. 2019 Nov 2;28(11):702-709. doi: 10.12968/jowc.2019.28.11.702. PMID 31721671
- [Background] Atkin L, Bucko Z, Conde Montero E, Cutting K, Moffatt C, Probst A, Romanelli M, Schultz GS, Tettelbach W. Implementing TIMERS: the race against hard-to-heal wounds. J Wound Care. 2019 Mar 1;23(Sup3a):S1-S50. doi: 10.12968/jowc.2019.28.Sup3a.S1. No abstract available. PMID 30835604
- [Background] Chamorro AM, Vidal Thomas MC, Mieras AS, Leiva A, Martinez MP, Hernandez Yeste MMS; Grupo UPP. Multicenter randomized controlled trial comparing the effectiveness and safety of hydrocellular and hydrocolloid dressings for treatment of category II pressure ulcers in patients at primary and long-term care institutions. Int J Nurs Stud. 2019 Jun;94:179-185. doi: 10.1016/j.ijnurstu.2019.03.021. Epub 2019 Apr 4. PMID 31048187
- [Background] Westby MJ, Dumville JC, Soares MO, Stubbs N, Norman G. Dressings and topical agents for treating pressure ulcers. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD011947. doi: 10.1002/14651858.CD011947.pub2. PMID 28639707
- [Background] Kim JY, Lee YJ. A study on the nursing knowledge, attitude, and performance towards pressure ulcer prevention among nurses in Korea long-term care facilities. Int Wound J. 2019 Mar;16 Suppl 1(Suppl 1):29-35. doi: 10.1111/iwj.13021. PMID 30793854
- [Background] Matsubara M, Banshodani M, Takahashi A, Kawai Y, Saiki T, Yamashita M, Shiraki N, Shintaku S, Moriishi M, Masaki T, Kawanishi H. Vascular access management after percutaneous transluminal angioplasty using a calcium alginate sheet: a randomized controlled trial. Nephrol Dial Transplant. 2019 Sep 1;34(9):1592-1596. doi: 10.1093/ndt/gfy143. PMID 29846686
- [Background] Stolt M, Hjerppe A, Hietanen H, Puukka P, Haavisto E. Local treatment of pressure ulcers in long-term care: a correlational cross-sectional study. J Wound Care. 2019 Jun 2;28(6):409-415. doi: 10.12968/jowc.2019.28.6.409. PMID 31166863
- [Result] Broussard KC, Powers JG. Wound dressings: selecting the most appropriate type. Am J Clin Dermatol. 2013 Dec;14(6):449-59. doi: 10.1007/s40257-013-0046-4. PMID 24062083
- [Result] Aljezawi M, Al Qadire M, Tubaishat A. Pressure ulcers in long-term care: a point prevalence study in Jordan. Br J Nurs. 2014 Mar 27-Apr 9;23(6):S4, S6, S8, S10-1. doi: 10.12968/bjon.2014.23.Sup6.S4. PMID 24690751